CLINICAL TRIAL: NCT03508791
Title: Effect of Patient Position on Arterial, End-tidal and Transcutaneous Carbon Dioxide Partial Pressure in Patients Undergoing Laparoscopic Surgery
Brief Title: Effect of Patient Position on Arterial, End-tidal and Transcutaneous Carbon Dioxide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201804-1
Record Dates: First submitted 2018-04-20; First posted 2018-04-26 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Ventilation Perfusion Mismatch
MeSH Terms: interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trendelenburg group (Active Comparator): Arterial, end-tidal, and transcutaneous carbon dioxide partial pressure are monitored in the Trendelenberg position
  Interventions: Other: Arterial carbon dioxide monitoring; Other: End-tidal carbon dioxide monitoring; Other: Transcutaneous carbon dioxide monitoring
- reverse Trendelenburg group (Active Comparator): Arterial, end-tidal, and transcutaneous carbon dioxide partial pressure are monitored in the reverse Trendelenberg position
  Interventions: Other: Arterial carbon dioxide monitoring; Other: End-tidal carbon dioxide monitoring; Other: Transcutaneous carbon dioxide monitoring

INTERVENTIONS:
Other: Arterial carbon dioxide monitoring — Arterial carbon dioxide partial pressure is monitored during the laparoscopic surgery undergoing in the Trendelenburg or reverse Trendelenburg positions.
Other: End-tidal carbon dioxide monitoring — End-tidal carbon dioxide partial pressure is monitored during the laparoscopic surgery undergoing in the Trendelenburg or reverse Trendelenburg positions.
Other: Transcutaneous carbon dioxide monitoring — Transcutaneous carbon dioxide partial pressure is monitored during the laparoscopic surgery undergoing in the Trendelenburg or reverse Trendelenburg positions.

SUMMARY:
Investigators evaluate the effect of patient position (Trendelenburg and reverse Trendelenburg) on arterial, end-tidal and transcutaneous carbon dioxide partial pressure in patients undergoing laparoscopic surgery.

DETAILED DESCRIPTION:
Investigators evaluate the effect of patient position (Trendelenburg and reverse Trendelenburg) on arterial, end-tidal and transcutaneous carbon dioxide partial pressure in patients undergoing laparoscopic surgery. Arterial carbon dioxide partial pressure is assessed intermittently before, during, and after pneumoperitoneum. End-tidal and transcutaneous carbon dioxide partial pressure are continuously monitored.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing laparoscopic surgery (expected duration of pneumoperitoneum > 1 hour) in the Trendelenburg or reverse Trendelenburg positions

Exclusion Criteria:

* hemodynamically unstable patients due to decompensated heart failure, sepsis, or symptomatic arrhythmia, etc.
* symptomatic pulmonary disease, chronic obstructive pulmonary disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-05-20 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Difference between arterial and end-tidal carbon dioxide pressures | baseline before CO2 pneumoperitoneum, every 30 minute during CO2 pneumoperitoneum, and 15 min after deflation of CO2
  Difference between arterial and end-tidal carbon dioxide partial pressures are calculated. (Arterial carbon dioxide partial pressure minus end-tidal carbon dioxide partial pressure)

SECONDARY OUTCOMES:
Agreement among arterial, end-tidal, and transcutaneous carbon dioxide partial pressure | baseline before CO2 pneumoperitoneum, every 30 minute during CO2 pneumoperitoneum, and 15 min after deflation of CO2
  Arterial, end-tidal, and transcutaneous carbon dioxide partial pressures are recorded and the agreement among the values is analyzed using the statistical test.